CLINICAL TRIAL: NCT02060695
Title: Temporal Relationship Between Motor Fluctuations and Nonmotor Fluctuations
Status: Recruiting | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, BS Jeon, Professor, Seoul National University Hospital
Other Study IDs: H-1109-081-378
Record Dates: First submitted 2014-02-03; First posted 2014-02-12 (Estimated); Last update posted 2017-05-03 (Actual); Status verified 2017-05

CONDITIONS: Parkinson Disease
Keywords: Parkinson disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to determine the temporal relationship between motor fluctuations and non-motor fluctuations in persons with Parkinson's disease.

Observational study case-only

DETAILED DESCRIPTION:
Objectives

1. how many patients will experience motor or nonmotor fluctuation during follow-up period?
2. in how many patients, does motor fluctuation precede nonmotor fluctuation?
3. in how many patients, does nonmotor fluctuation precede motor fluctuation?

Participants: persons with Parkinson disease in early stage who does not have motor or nonmotor fluctuation

Recruitment period: 3 years from the commencement of the study Follow-up period: 3 years for each participants

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of Parkinson disease by United Kingdom Parkinson's Disease Society Brain Bank criteria
* early stage

Exclusion Criteria:

* dementia (MMSE<26)
* persons who refuse participating

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: movement disorder clinic
Sampling Method: Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2012-09; Primary Completion 2030-06 (Estimated); Study Completion 2031-06 (Estimated)

PRIMARY OUTCOMES:
time period from the onset of disease to the occurrence of motor or nonmotor fluctuation | 6 months
  The proportion of participants with motor and/or nonmotor fluctuation will be evaluated at 6, 12, 18, 24, 30, and 36 months after the enrollment of each participant in order to determine the time course of motor/nonmotor fluctuation in persons with early stage of Parkinson's disease.

SECONDARY OUTCOMES:
sensitivity and specificity of self-diagnostic questionnaire of motor/nonmotor fluctuation | 3 years
  The participants will be checked regularly for the development of motor/nonmotor fluctuation during study period by both of self-diagnostic questionnaire and clinician. The validation of self-diagnostic questionnaire of motor/nonmotor fluctuation will be conducted compared to the clinician-evaluated occurrence of motor/nonmotor fluctuation.

OTHER OUTCOMES:
The proportion of participants with impulse control disorders | 6 months
  The presence of impulse control disorders including excessive shopping, binge eating, pathologic gambling, and hypersexuality will be checked with questionnaire at 6, 12, 18, 24, 30, and 36 months in order to determine the frequency of impulse control disorders among the participants
The proportion of participants with rapid eye movement (REM) sleep behavior disorder | 6 months
  The presence of REM sleep behavior disorder will be checked with questionnaire at 6, 12, 18, 24, 30, and 36 months in order to determine the frequency of REM sleep behavior disorder among the participants.
The proportion of participants with smoking history | 6 months
  The smoking history will be checked with questionnaire at 6, 12, 18, 24, 30, and 36 months in order to determine the influence of the smoking history to development of motor/nonmotor fluctuation.

CONTACTS AND LOCATIONS:
Overall Officials: Beom S Jeon, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Background] Witjas T, Kaphan E, Azulay JP, Blin O, Ceccaldi M, Pouget J, Poncet M, Cherif AA. Nonmotor fluctuations in Parkinson's disease: frequent and disabling. Neurology. 2002 Aug 13;59(3):408-13. doi: 10.1212/wnl.59.3.408. PMID 12177375
- [Background] Resnick RJ, Kole HK, Racker E. Multiple changes induced by cholera toxin contribute to the stimulation of aerobic lactate production in rat-1 fibroblasts. Arch Biochem Biophys. 1991 May 1;286(2):579-85. doi: 10.1016/0003-9861(91)90083-u. PMID 1654794
- [Background] Stacy M, Hauser R. Development of a Patient Questionnaire to facilitate recognition of motor and non-motor wearing-off in Parkinson's disease. J Neural Transm (Vienna). 2007 Feb;114(2):211-7. doi: 10.1007/s00702-006-0554-y. Epub 2006 Aug 10. PMID 16897594